CLINICAL TRIAL: NCT07171580
Title: TPD-REACH: Tailoring Post Discharge - Remote Education and Access for Cardiac Health
Brief Title: Tailoring Post Discharge - Remote Education and Access for Cardiac Health
Acronym: TPD-REACH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Responsible Party: Principal Investigator, Shuangbo Liu, Interventional Cardiologist, St. Boniface Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TPD-REACH Protocol
Record Dates: First submitted 2025-08-30; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction (MI)
Keywords: Percutaneous Coronary Intervention; Education; Support; Digital Health Tool; Remote Home Monitoring
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Comparing 3 interventional groups: 1) Standard Care 2) Education Only 3) Full Intervention (Education and Support)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care (SA) (No Intervention): Patients will receive standard education in hospital. They will not be registered in the RHM application or receive education modules, health care interviews or virtual appointments.
- Education Only (EA) (Experimental): Patients will be enrolled in the RHM application, allowing tracking of their access to the education modules. They will start with an introductory module, followed by one module per day for a total of 7 modules covering key topics related to ACS (Cardiac Rehabilitation, Heart Attack Risk Factors, Living with Heart Disease, Medications, Mental Health, Nutrition, Physical Activity). Participants that have atrial fibrillation will receive an additional education module on that topic, and participants with heart failure with receive an additional education module relating to that topic. Engagement for modules will be monitored, if any patient misses more than one module, they will be contacted for a reminder and troubleshooting. Participants will have access to the RHM education modules for 30 days post hospital discharge.
  Interventions: Other: Remote Home Monitoring - Education
- Full Intervention (Experimental): Patients will be enrolled in the RHM application. Patients will receive all interventions in the EA, and in addition, they will receive support through the RHM application. Patients will complete health care surveys three times a week, covering topics such as symptoms, vital signs, medication side effects, functional status, and whether they have questions or concerns. Patients will have three scheduled virtual appointments with a cardiologist on 1 day, 1 week, 2 weeks after discharge. If a patient misses a survey, they will be prompted. Patients will also have access to unscheduled health care interviews, virtual appointments, and a hotline for additional questions or concerns. Participants will have access to the RHM education modules and program support for 30 days post hospital discharge.
  Interventions: Other: Remote Home Monitoring - Education and Support

INTERVENTIONS:
Other: Remote Home Monitoring - Education — A virtual platform will be used to provide education to ACS patients post discharge.
  Arms: Education Only (EA)
Other: Remote Home Monitoring - Education and Support — A virtual platform will be used to provide education and support to ACS patients post discharge.
  Arms: Full Intervention

SUMMARY:
Heart attacks are one of the top causes of death in Canada, with over 2,100 cases treated each year in Manitoba. Even though hospital care has improved, the period after going home is still risky. Many patients feel anxious and unsure about their recovery, and without enough support, they often end up back in the emergency department (ED). This is an even bigger challenge for people in rural areas, where getting follow-up care can be much harder. Filling these gaps is important to help patients get better and to reduce stress on the healthcare system.

In a previous study, the investigators found that extra support made a big difference: only 8% of participants using a digital health tool returned to the ED within 30 days, compared to 22% of participants without it. Now, the investigators want to expand this study across Manitoba to see if digital health tools can help more people recover safely at home. The investigators will compare two types of follow-up care: education only versus education with extra support (like symptom tracking and virtual appointments). The investigators will look at how this affects hospital visits, mental well-being, and healthcare costs. The goal is to create a better support system for people after a heart attack, leading to healthier recoveries, less strain on hospitals, and better care for Manitobans - no matter where they live.

DETAILED DESCRIPTION:
STUDY AIM To evaluate the feasibility and effectiveness of a digital-based short-term post-discharge care program - providing education alone or with additional support - in reducing 30-day unexpected healthcare visits after discharge in low-to-intermediate risk ACS patients in Manitoba, compared to standard care.

STUDY OBJECTIVES Primary Objective: to compare the incidence of 30-day unexpected healthcare visits among low-intermediate risk ACS patients in Manitoba who receive education and support or education alone via a DHT, versus those receiving standard care.

Secondary Objectives: will examine 3 spheres of outcomes, across the 3 study groups:

1. Clinical Outcomes i. To examine and compare the occurrence of major adverse cardiovascular events (MACE) as a composite and individual components, including death, myocardial infarction (MI), repeat revascularization, readmission, stroke, vascular complications, or new HF requiring admission, at 30 days post-discharge ii. To explore the feasibility and acceptability of implementing a digital health platform intervention (DHPI) for extended short-term care for low-intermediate risk ACS patients in Manitoba at 30 days post-discharge iii. To identify patient-specific factors (e.g., home location, age, sex, gender) that may influence the effectiveness of the DHPI on healthcare utilization and recovery outcomes at 30 days post-discharge
2. Psychosocial Outcomes i. To evaluate patient-reported outcomes of mental health (e.g., anxiety, depression), quality of life, and satisfaction with care at 30 days post-discharge ii. To study the impact of the DHPI on patient activation measure, a marker of patients' knowledge, skills and confidence in self-managing their health at 30 days post-discharge iii. To assess patient satisfaction with the DHPI, focusing on usability, accessibility, and overall experience during recovery at 30 days post-discharge
3. Cost i. To conduct a cost-effectiveness analysis comparing the digital health platform interventions (education and support vs education alone) to standard care, examining healthcare resource utilization and potential cost savings at 30 days post-discharge

STUDY DESIGN This study is a single-center, pragmatic randomized controlled trial designed to evaluate post discharge support for low-intermediate risk ACS patients. Before hospital discharge, patients will be screened for eligibility. At discharge, eligible patients will be randomly assigned to one of three groups: (1) standard care; (2) education only and (3) education and support. The pragmatic design ensures that all study procedures-including recruitment, intervention, and follow-up-are closely integrated with routine clinical care, with minimal deviations beyond the study intervention itself. This approach enhances real-world applicability, making it easier to implement findings into everyday clinical practice. Study design and implementation are guided by the PRagmatic Explanatory Continuum Indicator Summary 2 (PRECIS-2) tool to ensure clinical relevance and feasibility. Full Research Ethics Board and institutional review board approval will be obtained before the study begins. The study will be registered on ClinicalTrials.gov.

STUDY INTERVENTION Remote Home Monitoring (RHM) is a secure, web-based, digital health application designed to support patients in their recovery. When used to its fullest extent, patients can access tailored education, real-time monitoring, track their health, and connect with care providers. RHM aims to improve patient knowledge, encourage self-management, and provide timely clinical support to reduce unexpected healthcare visits.

Study participants will be randomly assigned to one of three groups: standard care arm (SA), RHM education only arm (EA), RHM full intervention arm with education and support (FA). Before discharge, all patients will be provided with a blood pressure monitor and oximeter, allowing them to track their blood pressure and blood oxygen saturation at home. This not only supports ongoing health monitoring but also empowers patients to take an active role in managing their health.

(A) Standard Care Arm: Patients will receive standard education in hospital. They will not be registered in the RHM application or receive education modules, health care interviews or virtual appointments.

(B) Education Only Arm: Patients will be enrolled in the RHM application, allowing tracking of their access to the education modules. They will start with an introductory module, followed by one module per day for a total of 7 modules covering key topics related to ACS (Cardiac Rehabilitation, Heart Attack Risk Factors, Living with Heart Disease, Medications, Mental Health, Nutrition, Physical Activity). Participants that have atrial fibrillation will receive an additional education module on that topic, and participants with heart failure with receive an additional education module relating to that topic. Engagement for modules will be monitored, if any patient misses more than one module, they will be contacted for a reminder and troubleshooting. Participants will have access to the RHM education modules for 30 days post hospital discharge.

(C) Full Intervention Arm: Patients will be enrolled in the RHM application. Patients will receive all interventions in the EA, and in addition, they will receive support through the RHM application. Patients will complete health care surveys three times a week, covering topics such as symptoms, vital signs, medication side effects, functional status, and whether they have questions or concerns. Patients will have three scheduled virtual appointments with a cardiologist on 1 day, 1 week, 2 weeks after discharge. If a patient misses a survey, they will be prompted. Patients will also have access to unscheduled health care interviews, virtual appointments, and a hotline for additional questions or concerns. Participants will have access to the RHM education modules and program support for 30 days post hospital discharge.

Participants will be asked to complete questionnaires at three time points: baseline (link to access the questionnaires via REDCap will be sent on the day of hospital discharge), 14 days post discharge, and 30 days post discharge. These include validated tools to assess psychosocial well-being (GAD-7, PHQ-9, EQ-5D-5L, EQ-VAS) and patient activation (PAM-13). They will also complete surveys that cover demographics, health literacy, care transition, unexpected healthcare visits, and satisfaction with care. Responses will be securely collected and stored using REDCap, ensuring both convenience for participants and data integrity for analysis.

ELIGIBILITY:
Inclusion Criteria:

>18 years old, type 1 myocardial infarction27, resident of Manitoba

Exclusion Criteria:

Patients unable to consent or fully participate in the study due to:

1. Technology barriers

   1. Lack of digital device, internet access or data
   2. Discomfort with using technology
2. Communication or language barriers preventing participation
3. Cognitive or mental health limiting informed consent or participation

   1. Dementia or cognitive impairment
   2. Active or severe psychosis or other significant mental health conditions c. Active substance abuse
4. High-risk ACS where patients require more frequent or in person visits a. Cardiac:

   i. Coronary
   * Unrevascularizedleftmainormultivessellargeepicardialcoronary artery disease (>2.5mm)
   * Coronary artery bypass surgery (CABG) during index hospitalization ii. Arrhythmias
   * Cardiac arrest during index event/hospitalization (ventricular tachycardia (VT)/ventricular fibrillation (VF), pulseless electrical activity (PEA)) iii. Cardiomyopathy
   * Left ventricular ejection fraction (LVEF) <35% (most recent EF assessment)
   * Cardiogenic shock requiring pressors/inotropes for more than 24 hours
   * Requiring intubation/positive pressure ventilation/hi-flow oxygen for more than 24 hours
   * Switchedfromintravenous(IV)tooral(PO)loopdiureticwithinlast 48 hours
   * Change in PO loop diuretic dose within last 48 homes (home re- start of 80mg or less is allowed)
   * B-type natriuretic peptide (BNP) did not reduce by 30% iv. Cardiac Care Unit (CCU)/Intensive Care Unit (ICU) o Any CCU/ICU stay for more than 24 hours b. Medical: i. any condition with prognosis less than 1 year or a high LACE (Length of stay, Acuity of admission, Comorbidities, Emergency department use) score (>15)28 ii. any medical comorbidity requiring in-person assessment within 2 weeks TPD-REACH PROTOCOL v3 29Aug2025 8 of 17 TPD-REACH: Remote Education and Access for Cardiac Health iii. transition to an alternative living arrangement/compromised independent living iv. need medication adjustment or investigation within 2 weeks c. Social: i. severe financial strain ii. no fixed address or housing instability iii. severe food insecurity iv. significant hearing or vision impairment v. poor health literacy While we aim to promote health equity, patients facing these challenges need more support than this project can offer and should be connected to appropriate services before discharge.
5. Non-atherosclerotic causes of ACS (spontaneous coronary artery dissection, stress- induced cardiomyopathy, myocarditis) as the education and treatment is different
6. Any additional factor preventing full participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Unexpected Healthcare Visits | 30 days post hospital discharge
  30-day unexpected healthcare visits (including emergency department, urgent care, walk in clinic or nursing station)

SECONDARY OUTCOMES:
Composite of Events | 30 days post hospital discharge
  Composite of death, MI, repeat revascularization, readmission, stroke, vascular complication, new HF or needing admission
Individual Components of Composite Events | 30 days post hospital discharge
  Individual components of death, MI, repeat revascularization, readmission, stroke, vascular complication, new HF or needing admission
Individual Components of Composite Unexpected Healthcare Visits | 30 days post hospital discharge
  Individual components of unexpected healthcare visits including emergency department, urgent care, walk in clinic or nursing station
PAM-13 - Patient Activation Measure | Baseline (day of hospital discharge), 14 days post hospital discharge, and 30 days post hospital discharge
  This survey will measure patient knowledge, skills, and confidence in self- managing their health
Generalized Anxiety Disorder (GAD) - 7 | Baseline (day of hospital discharge), 14 days post hospital discharge, and 30 days post hospital discharge
  GAD-7 this survey measures self-report anxiety symptoms with a total score from 0-21. Lower scores indicate fewer anxiety symptoms
Patient Health Questionnaire (PHQ) - 9 | Baseline (day of hospital discharge), 14 days post hospital discharge, and 30 days post hospital discharge
  PHQ-9 this survey measures self-report depression symptoms with a total score from 0-27. Lower scores indicate fewer depressive symptoms
EQ-5D-5L - Health Related Quality of Life | Baseline (day of hospital discharge), 14 days post hospital discharge, and 30 days post hospital discharge
  EQ-5D-5L - This survey will measure 5 aspects of self-reported quality of life for patients. Each component is scored from 1-5 with a total score of the tool from 5-25. Lower scores indicate better outcomes
EQ-VAS - Health Related Quality of Life | Baseline (day of hospital discharge), 14 days post hospital discharge, and 30 days post hospital discharge
  EQ-VAS - this survey measures self-report quality of life on a scale of 0-100. Higher scores indicate better self reported quality of life
Patient Satisfaction Questionnaire | At 30 days post hospital discharge
  Patient Satisfaction with the care received and the study program
Overall Healthcare Cost Savings per Patient | 30 days post hospital discharge
  Average difference in healthcare costs between the study arms based on healthcare utilization.

CONTACTS AND LOCATIONS:
Locations (1):
- St Boniface Hospital, Winnipeg, Manitoba, Canada